CLINICAL TRIAL: NCT02168647
Title: The Blossom Project: "Be Well" Behavioral Wellness Study in Pregnancy to Prevent Excessive Gestational Weight Gain
Brief Title: The Blossom Project: "Be-Well" Behavioral Wellness Study in Pregnancy
Acronym: Be-Well
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, LBuckingham, Dr. Christina Campbell, Associate Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-199; 14-199 (Other: Iowa State University Institutional Review Board)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Excessive Weight Gain in Pregnancy With Baby Delivered
Keywords: Excessive gestational weight gain; Insulin resistance; Physical activity; Behavioral prenatal lifestyle intervention; Reduced carbohydrate intake; Self-determination theory; Motivational interviewing
MeSH Terms: conditions — Insulin Resistance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Lifestyle counseling (Experimental): Intervention group participants will take part in behavioral lifestyle counseling provided by a Registered Dietitian Nutritionist from week 14 of gestation through childbirth.
  Interventions: Behavioral: Behavioral Lifestyle counseling
- Control (Active Comparator): Participants in the control arm will receive no form of lifestyle intervention.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Behavioral Lifestyle counseling — Participants in the intervention group will take part in one-on-one visits with a registered dietitian nutritionist (RDN) from no later than week 14 to child birth at the OBGYN clinic where the participant receives her routine prenatal care or the Nutrition Wellness Research Center in the Iowa State Research Park. These visits will be coordinated with her routine prenatal appointment; therefore a minimum of 6 face-to-face meetings will occur. The counseling sessions will focus on appropriate weight gain during pregnancy through the use of an individualized meal plan, physical activity goals, and behavioral modification. Weight gain will be plotted on an IOM weight gain chart and discussed with study RDN.
  Arms: Behavioral Lifestyle counseling
Other: Control — Participants in the control arm will receive no form of lifestyle intervention. Women will be provided with usual care by their physician. Participants in the control arm will have their weight gain plotted on an IOM growth chart and sent electronically by research staff after each routine prenatal appointment. No other feedback on weight gain or behavior modification will be provided by the study RDN.
  Arms: Control

SUMMARY:
Multiple studies have demonstrated a very low prevalence of women meeting physical activity and weight gain recommendations during pregnancy. The aim of this study is to provide a lifestyle intervention to increase physical activity, reduce carbohydrate intake, prevent excessive gestational weight gain, decrease postpartum weight retention, and improve mental well-being compared to "usual care" using a randomized controlled design in pregnant women. Participants in the intervention group will receive behavioral lifestyle counseling and take part in monthly one-on-one visits with a registered dietitian (RDN) from approximately week 14 of their pregnancy to child birth. Participants in the "usual care" group (control) will not receive any lifestyle counseling. Data collected from this group will be used to compare the effectiveness of the lifestyle intervention. Unlike many studies examining diet and physical activity factors alone, this study evaluates additional psychosocial factors such as psychological health, self-efficacy, competence, motivation and barriers that may influence excessive gestational weight gain. In addition, the Self-Determination Theory framework will be used to measure how motivation and motivational interviewing strategies can help explain changes in volitional behavior.

DETAILED DESCRIPTION:
Pregnant women will be recruited using mass email recruitment, fliers posted at local community settings, and at local OBGYN offices in Ames,IA. Pregnant women will be recruited prior to their 14th week of gestation. Interested individuals will contact the Blossom Project staff for further information.

A randomized controlled design will be used. Following baseline data collection, women will be randomized into the intervention group (n=30) or control (n=30).

For this study, the goal is to have a total of 30 women in the intervention group and 30 in the control. With an attrition rate of 20% investigators plan to enroll 37 women per group. Furthermore, increased enrollment numbers will cover inconsistencies that may arise with missing or uninterpretable data.

Individuals who contact the Blossom Project will be screened for eligibility. Individuals that meet the inclusion and exclusion criteria will meet with a Blossom Project staff member to sign an informed consent form approved by the Iowa State University Institutional Review Board (ISU-IRB). A "medical consent form" (not the consent form for the study participant) will be sent to the woman's primary obstetric provider asking to confirm qualification criteria. Participants will then be asked to complete a medical history questionnaire.

Eligible participants will be asked to complete a maximum of four data collection periods. Participants will report to the Nutrition Wellness Research Center (NWRC) either on campus (HNSB 2021, 2022, 2023) or the facility located at 2325 North Loop Drive, Suite 6100, Ames, Iowa 50010, at the beginning and end of each of the four data collection periods. A "visit" or "data collection period" is defined as 8 days. There are 3 data collection periods during pregnancy (visits 1-3) and one post-partum visit (visit 4). Visit 4 is not an 8-day data collection period and will take no more than 90 minutes at the NWRC.

Data that will be collected during each of the data collection periods will include:

Visit 1: Prior to 14-weeks of pregnancy (8-14 weeks):

* Consent form: Participants will meet with a staff member to discuss the consent form and requirements of the study. Signed informed consent will be obtained from each participant.
* Medical provider consent: Medical providers will confirm qualification criteria for each participant. The medical provider consent must be received prior to a woman beginning the walking program (intervention group). Participants will sign this form at visit 1 to grant Blossom Project staff the permission to contact their medical provider.
* Medical history questionnaire: Each participant will fill out a medical history questionnaire.
* Physical activity assessment: Participants will receive verbal and written instructions on how to collect data regarding their physical activity. Each participant will wear 2 activity monitors to assess physical activity patterns over the 8-day monitoring period at weeks 8-14, 26-28 and 34-36 of their pregnancy. The sensors will be worn on the left arm over the triceps muscle (SenseWear Mini armband) and on the right leg over the quadriceps muscle (activPAL). All of these monitors have been used in our previous pregnancy studies with minimal complaints. Participants are required to record all their daily activities in a physical activity log that will be provided. The log is required to be recorded over the same consecutive 8 days for 24 hours a day that the 2 activity monitors are worn.
* Dietary assessment: Participants will receive verbal instructions on how to collect data regarding their dietary intake. Each woman will complete a 3-day weighed diet record which requires her to weigh and record all food and beverages consumed for 2 weekdays and 1 weekend day. Detailed written instructions will also be provided in a binder in a data collection bag with a dietary scale.
* Mental Well-being: Participants will complete the World Health Organization Quality of Life questionnaire that measures physical health, psychological health, social relationships and environment, the Edinburg Postnatal Depression Scale, which has been used for non-postnatal women as well as a screening scale for depression (pre-testing for our study), and a battery of standardized questionnaires regarding perceived self-efficacy, competence, motivation and barriers to control weight gain during pregnancy, and exercise safety beliefs. It should take approximately 15 minutes at each visit to complete these surveys.
* Anthropometric measurements: Height and weight will be measured. Body composition will be assessed using the BodPod, an air displacement plethysmograph that uses whole body densitometry to determine body composition using body mass and volume measures. We have used this technique in previous Blossom Project studies.
* Scheduling of follow-up appointment: Participants will schedule a time to return to the research facility the following week to return all monitors and materials (diet record, data collection bag, dietary scale).
* At enrollment, participants will fill out a Release of Medical Record form for their delivering hospital, to allow a Blossom Project staff member the ability to attain birth weight, birth length, head circumference, and APGAR scores at 1- and 5-minutes after the child is born utilizing medical records.

Visit 2 (weeks 26-28):

* Physical activity assessment via two monitors: SenseWear armband and the activPAL
* 3-day weighed diet record
* The same battery of the psychological variables (as described earlier) will be measured during this period. In addition a motivational interviewing fidelity checklist will be collected (through observations of the counseling sessions and self-reports from the counselor) to ensure that the motivational interviewing strategies were implemented.
* Anthropometric measurements: Weight 2-hour Oral Glucose Tolerance Test: The oral glucose tolerance test will consist of providing a fasted blood sample (following an overnight fast of 10-12 hours), consuming a 75-gram oral glucose solution and a blood sample at 60 minutes and 120 minutes following the consumption of the glucose solution. During this 2-hour period, the participant will be asked to remain seated at the research facility. The blood draw will be conducted by an experienced phlebotomist.

Visit 3 (weeks 34-36)

* Physical activity assessment via two monitors: SenseWear armband and the activPAL
* 3-day weighed diet record
* Measure of psychological variables (as described earlier) will be measured and a motivational fidelity checklist (as described in visit 2). During this visit, perceived support using the Health Care Climate questionnaire and psychological need satisfaction, using the Activity Feeling Scale, will be used to measure whether an autonomy supportive climate during the individualized lifestyle counseling was established for the intervention group.
* Anthropometric measurements: Weight

Visit 4 (2 months post-partum):

* Anthropometric measurements: Weight and maternal body composition using the BodPod.
* Infant Outcomes: birth outcomes; body composition using the PeaPod, air displacement plethysmograph used to assess infant body composition. The infant will be placed in a temperature-controlled test chamber of the PeaPod with a continuous outside air source for a brief amount of time (approximately one minute or less) while the measurement is taking place.
* Mental well-being: The Quality of Life scale, the postpartum depression scale and the perceived motivation and self-efficacy to continue to be physically active will be measured.

In order to protect the privacy of participants within the study records identifying participants will be kept confidential to the extent allowed by applicable laws and regulations. Records will not be made publicly available. To ensure confidentiality to the extent allowed by law, the following measures will be taken. Participants will be assigned a unique code that will be used on forms instead of their name. The signed consent form, medical provider consent form, and release of medical information forms will all need the woman's full name to identify her to her prenatal clinic and delivering hospital. These forms will be locked in a separate filing cabinet from the forms with the participant codes to prevent identification of the participants. If the results are published, the identity will remain confidential. The data obtained from the study will be regarded as privileged and confidential. The privacy will be maintained in any future analysis and/or presentation of the data with the use of coded identifications for each participant's data.Only members of the Blossom Project lab staff will have access to the data and study records. All data will be stored in a locked file cabinet with access only by the principal investigator and project staff. This data will be kept on hand in a separate locked file in the PI's laboratory (HNSB 1109, Iowa State University) until the results of the study have been published. Identifiers will be kept separate from the data. All electronic data is stored on a shared drive only accessible to the principal investigator and project staff which requires a password to access.

For statistical analysis data will be presented as descriptive variables. These variables will consist of diet, physical activity characteristics, adherence to daily step count recommendations, and postpartum outcomes. Between group differences, time effects, and corresponding interactions in the above variables will be assessed by a series of two-way analysis of variance contrasts. When identified, such differences will be further explored, in terms of relationships to the other measured characteristics of the study groups via correlations and regression-based modeling procedures. Statistical significance will be set at p < 0.05 and adjusted for any multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-45 with a pre-pregnancy BMI between 18.5-35.0 kg/m2 will be recruited for this study.
* Qualified pregnant women include those participating in a low-active or sedentary lifestyle defined as <3 30-minute exercise sessions per week and therefore, are not currently meeting physical activity guidelines during pregnancy.
* Participants will need to have qualification criteria confirmed by their medical provider prior to beginning the first data collection period.

Exclusion Criteria:

* Pregnant beyond 14 weeks gestation
* Multiple fetuses
* History of smoking during pregnancy
* History of gestational diabetes mellitus, pre-eclampsia, or chronic disease (e.g. Type 1 diabetes, Type 2 diabetes, heart disease, renal disease, or untreated thyroid conditions)
* Inability to comprehend the information shared during the informed consent process
* Any adverse reactions to armband monitors (e.g. metal allergies, electromagnetic devices)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Maternal Body Weight Change | From 14 weeks of gestation through 2 months post partum
  Gestational weight gain as measured by last pre-delivery weight minus self-reported pre-pregnancy weight.
  Maternal weight will be measured at each routine prenatal appointment and plotted on the IOM pregnancy weight gain chart.
  Body composition changes measured by BodPod at baseline and 2 months postpartum.

SECONDARY OUTCOMES:
Maternal Postpartum Depression and Perceived Quality of Life | Baseline through 2 months post partum
  World Health Organization Quality of Life questionnaire that measure physical health, psychological health, social relationships and environment.
  The Edinburg Postnatal Depression Scale
Maternal Insulin Resistance | Maternal 26th-28th week of gestation
  Plasma glucose concentrations and insulin resistance as measured from a oral glucose tolerance test.
Postpartum Weight Retention | From 14 weeks of gestation through 2 months post partum
  The difference between the weight at 2 months postpartum and the pre-pregnancy weight.

OTHER OUTCOMES:
Infant Outcomes | 2 months post partum
  Characteristics at birth including Apgar score, gestational age.
  Body composition (i.e. length, percent lean and fat mass) 2 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Campbell, Ph.D., Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

REFERENCES:
- [Derived] Buckingham-Schutt LM, Ellingson LD, Vazou S, Campbell CG. The Behavioral Wellness in Pregnancy study: a randomized controlled trial of a multi-component intervention to promote appropriate weight gain. Am J Clin Nutr. 2019 Apr 1;109(4):1071-1079. doi: 10.1093/ajcn/nqy359. PMID 30949691